CLINICAL TRIAL: NCT02923024
Title: Utilizing Existing Technology Using Patient Pings to Increase Physician Engagement at Oscar Health
Brief Title: Oscar Health Patient Pings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was cancelled before any participants were enrolled.
Sponsor: University of Pennsylvania (Other)
Collaborators: Oscar Health Insurance (Unknown)
Responsible Party: Principal Investigator, Amol Navathe, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 825856
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Emergency Room Utilization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): This arm will be usual care and there will be no intervention.
- Information (Experimental): In this arm, providers will be sent patient pings after a patient experiences a trigger event. The ping will be a fax sent from Oscar to the physician alerting them of an event their patient had.This trigger event could be an emergency room visit, admission to a hospital, or a hospital discharge event. The patient ping will be sent to the patient's doctor including primary care physicians and specialists. If the patient does not have a doctor, a ping will not be sent.
  Interventions: Behavioral: Patient Ping
- Information and Financial Incentives (Experimental): In this arm, providers will be sent patient pings after a patient experiences a trigger event. The ping will be a fax sent from Oscar to the physician alerting them of an event their patient had.This trigger event could be an emergency room visit, admission to a hospital, or a hospital discharge event. The patient ping will be sent to the patient's doctor including primary care physicians and specialists. If the patient does not have a doctor, a ping will not be sent. Physicians will be incentivized to see patients immediately via phone call or in office visit. Physicians receive a financial incentive for calling the member within 48 hours of trigger event and will receive a larger financial incentive for seeing the patient for an office visit within 7 days of trigger event.
  Interventions: Behavioral: Patient Ping

INTERVENTIONS:
Behavioral: Patient Ping — The patient ping will be a fax sent from Oscar Health to physician that will include information on the physician's patient's trigger event and contact information for the physician to reach out to the member.
  Arms: Information; Information and Financial Incentives

SUMMARY:
Oscar spends a significant amount of money every year on high cost high need individuals. With this increase in health care spending, Oscar Health is looking to expand care post emergency room and inpatient utilization for their members. In order to reduce hospital readmissions, reduce emergency room utilization, and increase the overall health of their members, Oscar is investing in a program to bring members better care through increased engagement with their primary care physician.

DETAILED DESCRIPTION:
Using their existing technology, Oscar is employing a randomized controlled trial among their physicians to improve their engagement and relationships with patients. The goal will be to test and refine patient pings as a provider engagement tool, with an eye toward using it within the broader approach to high-risk patients as well. The Penn team is helping to design the intervention, which includes helping with determining what the three arms will be and randomizing physicians and practice sites. They will implement a three-arm trial with the first arm being usual care (no pings), the second arm being the intervention of information, and the third arm being the intervention of information and financial incentives. In the two intervention groups, providers will be sent patient pings after a patient experiences a trigger event. This trigger event could be an emergency room visit, admission to a hospital, or a hospital discharge event. The patient ping will be sent to the patients doctors including primary care physicians and specialists. If the patient does not have a doctor, a ping will not be sent. In the third arm, physicians will be incentivized to see patients immediately via phone call or in office visit. Physicians will receive an incentive for calling the member within 48 hours of trigger event and will receive a larger financial incentive for seeing the patient for an office visit within 7 days of trigger event. This bonus payment will be paid to physicians uncoupled from usual reimbursement as a separate bonus check to increase salience. No pings will be sent to the physicians for the patients randomized to arm 1: usual care.

ELIGIBILITY:
Inclusion Criteria:

* Primary care and specialist physicians under contract with Oscar Health insurance

Exclusion Criteria:

* Any primary care and specialist physician not under contract with Oscar Health.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Patient office visits with physician | Within 7 days of trigger event and patient ping
  The study team will measure the number of patients that saw their physician within seven days of the trigger event and patient ping.
Physician phone call to patient | 48 hours of trigger event and patient ping
  The study team will measure the number of patients that received a phone call from their physician within 48 hours of trigger event.

SECONDARY OUTCOMES:
Number of emergency room visits post trigger event | 6 months
  The study team will measure emergency room utilization post trigger event.
Number of outpatient visits post trigger event | 6 months
  The study team will measure outpatient utilization post trigger event.

IPD SHARING:
Plan to Share IPD: No